CLINICAL TRIAL: NCT03586531
Title: Renal Biopsy Findings In Patients With Unexplained Elevated Serum Creatinine In Assiut University Hospital
Brief Title: Renal Biopsy Unexplained Elevated Serum Creatinine
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Radwa Ellisy, Principal investigator, Assiut University
Other Study IDs: RBUESCAUH
Record Dates: First submitted 2018-06-19; First posted 2018-07-13 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Renal Impairment
Keywords: renal biopsy, CKDu Egypt, unexplained elevated serum creatinine
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Renal biopsy spicemin retained in diluted formaldyde
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: renal biopsy — Renal biopsy samples will be obtained by a percutaneous method using a spring-loaded Trucut® biopsy needle under real time ultrasound guidance. Biopsy samples will be processed for light microscopy with special staining will be done: Schiff periodic acid, Masson trichrome and methenamine silver.and immunofluorescence studies to evaluate IgA, IgG, IgM, complement C1q and C3, fibrin, and kappa and lambda light chain deposits.

SUMMARY:
Patients presented with unexplained elevated serum creatinine including vast varieties of acute or chronic kidney disease. Renal biopsy may include acute and chronic interstitial nephritis, glomerulosclerosis and tubular atrophy, acute tubular necrosis, rapidly progressive glomerulonephritis, granulomatous glomerulonephritis, monoclonal gammopathy, myeloma kidney or thrombotic microangiopathy .

Renal biopsy definitely still plays the most vital and irreplaceable role in the investigations of cases with unexplained renal impairment. Despite a vastly variable biopsy results between patients, renal biopsy has helped in determining the best treatment and prognosis for the patients.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) can be considered to be present if a patient has a glomerular filtration rate (GFR) <60 mL/min or markers of structural kidney disease that have been present for >3 months. These include proteinuria, haematuria and radiological abnormalities.

CKD is an important global-health challenge. It is found in 10% of the global population. The age-standardized global prevalence of CKD stages 1-5 in adults aged 20 and older was 10.4% in men and 11.8% in women. The incidence of end-stage renal failure is increasing worldwide with an annual growth rate of 8%.

In 2010, the total number of renal replacement therapy (RRT) patients worldwide amounted to 2.6 million, whereas the number of patients needing this treatment was estimated to be between 4.9 and 9.7 million, with the largest gap between need and supply of RRT in low-income countries, particularly in Asia and Africa.

In 2013, Egypt was among the countries for which CKD was ranked in the top 10 for years of life lost (YLL, calculated by multiplying numbers of deaths by life expectancy at time of death in a reference population) due to premature death and disability-adjusted life years (DALYs) to reflect the degree of disability such as pain or functional limitations caused by each condition.

Early detection and treatment of CKD can be implemented at minimal cost and will reduce the burden of ESRD, improve outcomes of diabetes and cardiovascular disease (including hypertension), and substantially reduce morbidity and mortality from non communicable diseases (NCDs).

Diabetes and hypertension are the predominant risk factors for chronic kidney disease (CKD) globally. Infectious diseases resulting in glomerulonephritis are also important in low-income countries. However, in the past two decades, a severe form of CKD has been reported in individuals without these risk factors. CKD of unknown etiology (CKDu) affects adults in their third to fifth decade and is often fatal due to disease progression and lack of dialysis or transplant options in the involved geographic areas. CKDu has been reported in Sri Lanka, several Central American countries, the state of Andhra Prakesh in India and Egypt.

Besides the conventional work up of CKD cases, renal biopsy is indicated in patients with CKD whose kidneys are normal or near normal in size, where the diagnosis cannot be made by other means.

Renal biopsy definitely still plays the most vital and irreplaceable role in the investigations of cases with unexplained renal impairment. Despite a vastly variable biopsy results between patients, renal biopsy has helped in determining the best treatment and prognosis for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Impaired renal function (serum creatinine> 115umol/l serum urea > 8 mmol/l)
* Negative immunological markers i.e ANA, ANCA, cryoglobulin, and complement level.

Exclusion Criteria:

* Diabetic patients.
* Hypertensive patients.
* All causes of Acute kidney injury
* Bleeding diathesis.
* Known cases of primary or secondary glomerulonephritis.
* Patients with a single functioning kidney
* small sized kidneys
* Multiple renal cysts and ADPKD.
* Patients with asymmetrical kidney size.
* Patient with active infections.
* HBsAg, HCV and HIV positive patients.
* Obstructive uropathy.
* Patients with active malignancies e.g multiple myeloma
* Renal transplant.
* Refusal to do a biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients attended to outpatient clinics or admitted to internal medicine department in assiut univesity hospital
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
correlation between histopathological findings and serum creatinine in umol/l | 3 years
  histopathological patterns in term of glomerlular pathology, interstitial fibrosis, tubular injury and serum creatinine in umol /l

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Derived] Ellisy RA, Tony EA, Ismail W, Radi R, Seddik MI, Abdel Aziz EM. Clinicopathological characteristics and outcomes of patients with unexplained renal impairment: A single center study. Nefrologia (Engl Ed). 2025 Mar;45(3):249-258. doi: 10.1016/j.nefroe.2025.02.012. PMID 40082054